CLINICAL TRIAL: NCT05233033
Title: A Phase 1, Multicenter, Open-Label, Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, PK/PD, and Clinical Activity of Intravenously Administered KT-413 in Adult Patients with Relapsed or Refractory B-cell NHL
Brief Title: Safety, PK/PD, and Clinical Activity of KT-413 in Adult Patients with Relapsed or Refractory B-cell NHL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kymera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KT413-DL-101
Record Dates: First submitted 2022-01-18; First posted 2022-02-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Non Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma; DLBCL; MYD88 Gene Mutation
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1a Dose Escalation (Experimental)
  Interventions: Drug: KT-413
- Phase 1b Dose Expansion MYD88MT (Experimental): KT-413 given at the RP2D identified in Phase 1a Dose Escalation in patients with MYD88 mutant DLBCL.
  Interventions: Drug: KT-413
- Phase 1b Dose Expansion MYD88WT (Experimental): KT-413 given at the RP2D identified in Phase 1a Dose Escalation in patients with MYD88 wild type DLBCL.
  Interventions: Drug: KT-413

INTERVENTIONS:
Drug: KT-413 — KT-413 will be supplied as 10mg/mL concentration frozen solution to be administered intravenously per the protocol defined dose level.

SUMMARY:
This Phase 1a/1b study will evaluate the safety, tolerability and the pharmacokinetics/ pharmacodynamics (PK/ PD) of KT-413 in patients with R/R NHL. The Phase 1a stage of the study will explore escalating doses of single-agent KT-413. The Phase 1b stage will be split into 2 expansion cohorts to further characterize the safety, tolerability and the pharmacokinetics/ pharmacodynamics (PK/ PD) of KT-413 in MYD88 mutant and MYD88 wild-type R/R DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1a Only:

  * Histologically confirmed diagnosis of B-cell NHL according to the 2016 World Health Organization (WHO) classification. Diffuse large B-cell lymphoma (DLBCL) includes: DLBCL not otherwise specified (NOS) with or without MYC and BCL2 and/or BCL6 rearrangements; Epstein-Barr virus (EBV) positive DLBCL, NOS; human herpesvirus 8 (HHV8) positive DLBCL, NOS; DLBCL associated with chronic inflammation; and Primary cutaneous DLBCL, leg type. Patients with indolent lymphoma are eligible if they meet criteria for systemic treatment.
  * Clinicopathological diagnosis of Waldenström's Macroglobulinemia (WM) based on the consensus panel criteria from the Second International Workshop on WM
  * Histologically/cytologically confirmed relapsed/refractory Primary Central Nervous System Lymphoma (PCNSL) by cerebrospinal fluid (CSF) or biopsy. PCNSL patients are considered eligible if the Investigator believes that there is no other reasonable treatment alternative.

    * Note: Patients with HIV-associated PCNSL are not eligible.
    * Note: Patients with secondary CNS metastases are eligible assuming they meet other study criteria. Patients with secondary CNS metastases include those who have synchronous systemic and CNS involvement or those who have been previously treated and relapsed with isolated CNS involvement.
* Phase 1b Only: Histologically confirmed diagnosis of DLBCL according to the 2016 WHO classification including: DLBCL not otherwise specified (NOS) with or without MYC and BCL2 and/or BCL6 rearrangements; Epstein-Barr virus (EBV) positive DLBCL, NOS; HHV8+ DLBCL, NOS; DLBCL associated with chronic inflammation; and Primary cutaneous DLBCL, leg type.
* Disease relapsed and/or refractory to at least 2 accepted standard systemic regimens for all indications except PCNSL. For PCNSL, patients must be relapsed and/or refractory to at least 1 prior regimen.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 at Screening.
* Adequate organ and bone marrow function, in the absence of growth factors
* Patients of child-bearing potential must use adequate contraceptive measures to avoid pregnancy for the duration of the study as defined in the protocol

Exclusion Criteria:

* Infection with hepatitis B (HBV), hepatitis C (HCV), or active viral infection with human immunodeficiency virus (HIV).
* Radiation treatment within 4 weeks prior to first dose of study drug, unless the tumor site continues to increase in size after the patient has completed radiotherapy treatment.
* Major surgery requiring general anesthesia within 4 weeks prior to first dose of study drug, unless the tumor site continues to increase in size after the patient has completed radiotherapy treatment.
* Ongoing unstable cardiovascular function including history of myocardial infarction within 3 months of planned start of study drug.
* Patient has not recovered from any clinically significant AEs of previous treatments to pre-treatment baseline or Grade 1 prior to first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
To establish the Maximum Tolerated Dose (MTD) | Within first 3 weeks of treatment
  Phase 1a
Number of Participants with protocol specified Dose Limiting Toxicities (DLTs) | Within first 3 weeks of treatment
  Phase 1a
Dose recommended for future studies | Within first 3 weeks of treatment
  Phase 1a/1b
Clinical Laboratory Abnormalities | Clinical laboratory abnormalities will be assessed from the time ICF signature through 30 days post dose or prior to start of a new anticancer therapy
  Incidence and severity of clinical laboratory abnormalities in serum chemistry, hematology, coagulation parameters, and urinalysis tests as assessed by CTCAE v5.0 (Phase 1a/1b)
Adverse Event Parameters | Adverse Event Parameters will be assessed from the time ICF signature through 30 days post dose or prior to start of a new anticancer therapy
  Incidence and severity of adverse events as assessed by CTCAE v5.0 (Phase 1a/1b)
ECG Parameters | ECG Parameters will be assessed from the time ICF signature through 30 days post dose or prior to start of a new anticancer therapy
  Changes in the ECG parameters, including heart rate and measures PR, QRS, QT, and QTc intervals as assessed by CTCAE v5.0 Phase 1a/1b

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve for KT-413 from time zero to last quantifiable time point (AUC0-t) | Blood samples for PK analysis collected at multiple visits during cycle 1 and cycle 2 (each cycle is 21 days)
  Phase 1a/1b
Maximum Plasma Concentration of KT-413 (Cmax) | Blood samples for PK analysis collected at multiple visits during cycle 1 and cycle 2 (each cycle is 21 days)
  Phase 1a/1b
Time of maximum plasma concentration of KT-413 (Tmax) | Blood samples for PK analysis collected at multiple visits during cycle 1 and cycle 2 (each cycle is 21 days)
  Phase 1a/1b
Half-life of KT-413 [if data permits (T1/2)] | Blood samples for PK analysis collected at multiple visits during cycle 1 and cycle 2 (each cycle is 21 days)
  Phase 1a/1b
Amount of KT-413 excreted in urine from time zero to last collected timepoint (Ae0-t) | Urine samples for PK analysis collected during the first cycle (21 day cycle)
  Phase 1a/1b
Evidence of clinical activity of KT-413 as determined by Objective Response Rate (ORR) | From date of baseline scan until the date of first documented progression or date of death from any cause, whichever came first, about 18 months
  Phase 1a/1b
Duration of Response (DOR) as assessed by the Investigator | From date of baseline scan until the date of first documented progression or date of death from any cause, whichever came first, about 18 months
  Phase 1a/1b
Progression-free survival (PFS) as assessed by the Investigator | From time of entry on study through progression, up to 18 months
  Phase 1b
Disease Control Rate (DCR) as assessed by the investigator | From date of baseline scan until the date of first documented progression or date of death from any cause, whichever came first, about 18 months
  Phase 1b
Overall Survival (OS) as assessed by the investigator | From time of entry on study through death or date last known alive at end of follow-up, up to 18 months
  Phase 1b

OTHER OUTCOMES:
KT-413 levels in peripheral blood mononuclear cells | Blood samples for PD analysis collected at multiple visits during cycle 1 and cycle 2 (each cycle is 21 days)
  Phase 1a/1b

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Gollerkeri, MD, Study Director — Kymera Therapeutics, Inc.
Locations (8):
- United States (6):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Norton Cancer Institute, Louisville, Kentucky
  - Henry Ford Health System, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
- United Kingdom (2):
  - University College London Hospitals, London
  - University Hospital Southampton NHS Foundation Trust, Southampton